CLINICAL TRIAL: NCT04919460
Title: Research on Optimization and Evaluation of Oral Cancer Screening Methods
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CN-oral
Record Dates: First submitted 2021-05-27; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Oral Cancer
Keywords: Oral cancer; Screening Method
MeSH Terms: conditions — Mouth Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clinical observation combined with pathological biopsy (Other): Clinical observation (including inspection and palpation) combined with pathological biopsy. That is, inspecting and palpating the oral cavity and neck of the screened object. If positive lesions are found, then further pathological biopsy will be performed.
  Interventions: Other: clinical observation combined with pathological biopsy
- Clinical observation, in vivo staining combined with pathological biopsy (Experimental): Clinical observation (including inspection and palpation), in vivo staining (reagent: toluidine blue) combined with pathological biopsy. That is, inspecting and palpating the oral cavity and neck of the screened object. At the same time, in vivo staining is performed on each participant. The reagent used for staining is toluidine blue. As long as the screening subjects found positive lesions or abnormal living body staining, pathological biopsy was performed.
  Interventions: Other: Clinical observation, in vivo staining (reagent: toluidine blue) combined with pathological biopsy

INTERVENTIONS:
Other: clinical observation combined with pathological biopsy — Inspecting and palpating the oral cavity and neck of the screened object. If positive lesions are found, then further pathological biopsy will be performed.
  Arms: clinical observation combined with pathological biopsy
Other: Clinical observation, in vivo staining (reagent: toluidine blue) combined with pathological biopsy — (2) Inspecting and palpating the oral cavity and neck of the screened object. At the same time, in vivo staining is performed on each participant. The reagent used for staining is toluidine blue. As long as the screening subjects found positive lesions or abnormal living body staining, pathological biopsy was performed.
  Arms: Clinical observation, in vivo staining combined with pathological biopsy

SUMMARY:
An evaluation and validation study on oral cancer screening methods will be carried out, and two different methods will be used for oral cancer screening among the population. The two different methods are: (1) clinical observation (including inspection and palpation) combined with pathological biopsy. (2) Clinical observation (including inspection and palpation), in vivo staining (toluidine blue) combined with pathological biopsy. By evaluating and comparing the sensitivity and specificity of the two screening methods, the more effective oral cancer screening method will be selected.

DETAILED DESCRIPTION:
An evaluation and validation study on oral cancer screening methods will be carried out, and two different methods will be used for oral cancer screening among the population. The two different methods are: (1) clinical observation (including inspection and palpation) combined with pathological biopsy. That is, inspecting and palpating the oral cavity and neck of the screened object. If positive lesions are found, then further pathological biopsy will be performed. This is also the commonly used screening method for oral cancer now; (2) Clinical observation (including inspection and palpation), in vivo staining (toluidine blue) combined with pathological biopsy. That is, toluidine blue staining is performed at the same time as the inspection and palpation of the oral cavity and neck of the screening object. As long as the screening subjects found positive lesions or abnormal living body staining, pathological biopsy was performed. By evaluating and comparing the sensitivity and specificity of the two screening methods, the more effective oral cancer screening method will be selected. Finally, we will carry out prospective controlled population studies in high-risk areas and non-high-risk areas to further evaluate the effectiveness and feasibility of screening method after selection.

ELIGIBILITY:
Inclusion Criteria:

* aged 40-69 years old.

Exclusion Criteria:

* No.

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The rate of participants being detected as positive | 1 year
  Among all participants, the rate of being tested positive by two methods

IPD SHARING:
Plan to Share IPD: Undecided